CLINICAL TRIAL: NCT02910622
Title: Pilot Study Evaluating the Oncogramme: Analysis of Response to Induction Treatment of Patients With Breast or Ovarian Cancer.
Acronym: ONCO S-O
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I09018 (ONCOGRAMME S-O)
Record Dates: First submitted 2016-09-12; First posted 2016-09-22 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: breast; ovarian; cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor fragment
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Oncogramme breast: Taking a fragment of breast tumors taken from a specimen. Cells fragment are cultured for 7 days. The effects of chemotherapy are studied on these cells through chimio-oncogramme
  Interventions: Other: Chimio-oncogramme
- Oncogramme ovarian: Taking a fragment of ovarian tumors taken from a specimen. Cells fragment are cultured for 7 days. The effects of chemotherapy are studied on these cells through chimio-oncogramme
  Interventions: Other: Chimio-oncogramme

INTERVENTIONS:
Other: Chimio-oncogramme — Cells fragment are cultured for 7 days. The effects of chemotherapy are studied on these cells through chimio-oncogramme.

SUMMARY:
The choice of treatments for cancers by systemic way - chemotherapy, hormone therapy and targeted therapies - is currently defined by criteria for population groups and not to an individual. These expensive treatments - in financial terms and quality of life - will be effective for some and administered unnecessarily for other because there is no predictive test of response for a given individual.

For breast cancer, the usual treatment includes the first surgery and adjuvant therapies (chemotherapy, hormonal therapy ...) whose effectiveness will be assessed after many years as the occurrence or not of a recurrence or metastases.

These systemic treatments can also be administered before surgery to reduce the tumor volume and secondarily allow less mutilating surgery: it is the principle of treatment neo adjuvant. In this case, the efficiency will be evaluated more quickly.

In practice, a patient with breast cancer suspicion has a biopsy which confirms the diagnosis and defined the parameters (hormone receptors, cytological grade, receptor monoclonal antibodies ...) that guide to the most appropriate type of treatment.

Tumor size is evaluated in neo adjuvant pre-treatment by imaging: mammography, ultrasound and MRI.

At the end of this medication, the evaluation of the response is achieved by radiology and surgery.

Pathological examination evaluates and precise response by the criteria of Chevallier and / or Sataloff. An ex vivo test for predicting the response of cells to different chemotherapy regimens, the oncogramme, was developed by Oncomedics, a young company whose technology is derived from the University of Limoges.

Clinical response and / or histopathological could be compared in a reasonable time (2-6 months), the results of the oncogramme proposed by Oncomedics whether the efficiency obtained in vivo is that predicted by the ex vivo test.

It is the same in the metastatic setting when there is an available target for biopsy and assessment of response.

The management of ovarian cancer in advanced stages can also benefit from a radiological and histopathological evaluation strategy before and after systemic treatment to compare the in vivo results with those predicted by ex vivo by Oncomedics.

DETAILED DESCRIPTION:
A fragment of Breast/Ovarian tumors will be taken from a specimen or a cold biopsy, tissue from patients diagnosed with breast cancer or ovarian cancer before starting an induction treatment stage IIIc and IV pleural IFGO operable.

* Culturing the cells obtained from the tumor fragment by Oncomedics in a defined medium and provided for enriching tumor cells compared to stromal cells.
* Maintaining the cells in culture for 7 days.
* Effects of conventional chemotherapy (corresponding to protocols) on these cells for 72 hours (growth chambers) by Oncomedics (chimio-oncogramme).
* For each chemotherapy tested, measuring the proportion of dead cells / total cells.
* Retained by Oncomedics results, not given to the nursing team. The patient will be treated and followed up in the usual way.
* At the end of the study, comparing the in vitro results (chimio-oncogramme) to the patient response to the same chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years.
* Patient with breast cancer needed starting an induction therapy or neo-adjuvant or metastatic but inoperable position (isolated bone metastases, skin permeation nodule).
* Patient Diagnosed with ovarian cancer before starting an induction treatment stage IIIc and IV pleural IFGO operable.
* Measurable disease according to RECIST 1.1 criteria by Magnetic resonance imaging (MRI), tomodensitometry scan or assessable by positron emission tomography scan (PET-SCAN) according to European Organisation for Research and Treatment of Cancer (EORTC) or Chevallier criteria and / or Sataloff post-neo adjuvant for breast or assessable during surgery for carcinomatosis by score Sugarbaker
* Patient has not expressed opposition to the use of their residual tumor
* Lack of cancer within 5 years with the exception of basal cell carcinoma or squamous cell cancer or in situ cervix Treaty
* Patients not included in a therapeutic trial with an experimental molecule in the indication concerned.

Exclusion Criteria:

* Lack of contraception for women of childbearing age
* Use of targeted therapy, hormone therapy, radiation therapy concomitantly
* Inability to submit to monitoring for geographical, social or psychological reasons
* Nobody deprived of liberty by administrative or judicial decision or person under guardianship.
* Difficulty understanding of the Protocol
* Social uninsured patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with breast cancer needed starting an induction therapy neo-adjuvant or metastatic but inoperable position (isolated bone metastases, skin permeation nodule). And patient diagnosed with ovarian cancer before starting an induction treatment stage IIIc and IV pleural IFGO (International federation of gynecology obstetric) operable.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
In vitro analysis of chemotherapy responses | Days 7
  Evaluate the predictive value of chemo-oncogramme on the patients response to the same (s) chemotherapy (s)

SECONDARY OUTCOMES:
Radiological Evaluation of the in vivo response | Days 7
  Radiological Evaluation of the in vivo response by RECIST or EORTC criteria

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University Hospital, Bordeaux
  - University Hospital, Limoges

IPD SHARING:
Plan to Share IPD: No